CLINICAL TRIAL: NCT00601861
Title: A Single Arm, Single-centre, Open-label, Exploratory Trial of Recombinant Interleukin-21 Administered Subcutaneously for 4 Weeks as Neo-adjuvant Treatment Prior to Sentinel Lymph Node/Complete Lymph Node Dissection Followed by 8 Weeks of Adjuvant Treatment in Subjects With Stage III Malignant Melanoma
Brief Title: Effect of rIL-21 on Metastases in Lymph Nodes in Melanoma Skin Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: See termination reason in detailed description
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NN028-1801; 2006-005350-79 (EudraCT Number)
Record Dates: First submitted 2008-01-03; First posted 2008-01-28 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2017-02

CONDITIONS: Cancer; Malignant Melanoma
MeSH Terms: conditions — Neoplasms; Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Drug: recombinant interleukin-21

INTERVENTIONS:
Drug: recombinant interleukin-21 — Fixed and equal dose for s.c. injection, 3 times weekly
  Other Names: rIL-21, NN028

SUMMARY:
The trial is conducted in Europe. This trial aims for a comparison of the pathology in lymph nodes before and after the effect of recombinant interleukin-21 in patients with stage III melanoma

DETAILED DESCRIPTION:
The decision to discontinue the NN028-1801 trial is not due to any safety concerns. The trial was terminated as a result of a strategic decision by the sponsoring company.

ELIGIBILITY:
Inclusion Criteria:

* Stage III melanoma
* ECOG performance status 0-1

Exclusion Criteria:

* Signs of stage IV melanoma
* Safety variables

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2008-02-13 (Actual); Primary Completion 2008-06-25 (Actual); Study Completion 2008-06-25 (Actual)

PRIMARY OUTCOMES:
Complete pathological response rate in the lymph nodes | After 4 weeks of treatment

SECONDARY OUTCOMES:
Safety | For the duration of the trial
Immunomodulatory effects | For the duration of the trial
Relapse free survival | For up to 4 years after the final visit or until progression of the disease in order to assess the relapse free survival (RFS)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Berlin, Germany

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com